CLINICAL TRIAL: NCT03196453
Title: Sopusuhtainen Lapsi - Kliininen Tutkimus Painonhallinnasta
Brief Title: Fit Child - Clinical Study on Weight Control
Acronym: FITCHI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study protocol has been applied in a new study, after te COVID. New registration.
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Erika Isolauri, Professori, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T6161/2017
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2017-06

CONDITIONS: Overweight; Nutrition Disorder, Child; Weight Change, Body
Keywords: overweight; probiotic; weight management
MeSH Terms: conditions — Overweight; Child Nutrition Disorders; Body Weight Changes | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: double blind, placebo controlled,
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Probiotic (Active Comparator): Lactobacillus rhamnosus GG
  Interventions: Dietary Supplement: Probiotic
- Probiotic and protein (Active Comparator): Lactobacillus rhamnosus GG and whey protein isolate
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — probiotic and/or placebo intervention in toddlers
  Other Names: FITCHI (Fit Child)

SUMMARY:
Children with abnormal weight development of BMI will be given either placebo or a probiotic protein formula and measures of weigh gain during a 3-mont treatment will be conducted

DETAILED DESCRIPTION:
In this study, children with abnormal weight development of BMI will be recruited and the gut microbiota will be modified using one of there treatment schedules. The subjects will be divided into three groups 1) receiving a daily drink with protein drink with a probiotic Lactobacillus rhamnosus GG or 2) placebo drink and/or 3) drink with Lactobacillus rhamnosus GG.

The children will give a faecal sample in the beginning and at the end and similarly also a blood sample. The faecal sample will be used for analysis of microbiota and differences in microbiota between the groups. Blood samples will be analysed for obesity related biomarkers.

Body weight is followed at home and at frequent intervals of the study and analyses made for overweight related biomarkers.

ELIGIBILITY:
Inclusion Criteria: 2-5 year old child with early weight gain and abnormal BMI, parental concern on weight gain/development

-

Exclusion Criteria:Medicines influencing gastric or intestinal function, antibiotic treatment during the last 6 months, use of specific probiotics

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-05-25 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
weight gain | 3 months
  body weight

SECONDARY OUTCOMES:
Blood biomarkers | 3 months
  Subar
Weight change | 3 months
  Weight change

CONTACTS AND LOCATIONS:
Overall Officials: Erika Isolauri, Principal Investigator — University of Turku, Department of Pediatrics
Locations (1):
- University of Turku and University Hospital Turku, Turku, Varsinaissuomi, Finland

IPD SHARING:
Plan to Share IPD: No
IPD will be shared once the study has been completed and analysed